CLINICAL TRIAL: NCT06041152
Title: Does Psilocybin Change Synaptic Density in the Brains of Patients With Amnestic Mild Cognitive Impairment
Brief Title: Does Psilocybin Change Synaptic Density in Amnestic Mild Cognitive Impairment
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Philip Gerretsen, Clinician Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 101-2021
Record Dates: First submitted 2023-08-01; First posted 2023-09-18 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Amnestic Mild Cognitive Impairment
Keywords: amnestic mild cognitive impairment; psilocybin; SV2A; positron emission tomography; synaptic vesicular density
MeSH Terms: interventions — Psilocybin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Amnestic Mild Cognitive Impairment Participants Receiving Psilocybin (Experimental): Receiving 2 doses of 25mg of psilocybin separated by 1 week.
  Interventions: Drug: Psilocybin
- Healthy Participants Receiving Psilocybin (Experimental): Receiving 2 doses of 25mg of psilocybin separated by 1 week.
  Interventions: Drug: Psilocybin
- Amnestic Mild Cognitive Impairment Participants Receiving Placebo (Placebo Comparator): Receiving 2 doses of placebo separated by 1 week.
  Interventions: Drug: Placebo
- Healthy Participants Receiving Placebo (Placebo Comparator): Receiving 2 doses of placebo separated by 1 week.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Psilocybin — 2 macrodoses of 25mg separated by one week.
  Arms: Amnestic Mild Cognitive Impairment Participants Receiving Psilocybin; Healthy Participants Receiving Psilocybin
Drug: Placebo — 2 doses of placebo separated by one week.
  Arms: Amnestic Mild Cognitive Impairment Participants Receiving Placebo; Healthy Participants Receiving Placebo

SUMMARY:
The goal of this clinical trial is to investigate the effects of psilocybin on synaptic vesicular density (SVD) as measured by the positron emission tomography (PET) radiotracer, 18F-SynVesT-1, in participants with amnestic Mild Cognitive Impairment (aMCI) and healthy participants. The investigators hypothesize that SVD levels in the brain will be higher following the ingestion of psilocybin in comparison to placebo, and that increases in SVD will be associated with improvements in cognition.

60 participants (30 with aMCI, and 30 sex and age matched healthy volunteers) will:

* Be randomized to receive either:

  1. Two 25 mg macrodoses of psilocybin separated by 1 week.
  2. Two placebo doses separated by 1 week.
* Receive a baseline 18F-SynVesT-1 PET scan, clinical, and neuropsychological assessments.
* Receive a 18F-SynVesT-1 PET scan one week after the last dose of treatment.
* Receive a third PET scan at any time within 4 weeks of the screening visit to quantify tauopathy with the [18F]T807 radiotracer.
* Receive clinical and neuropsychological testing 1, 4, and 12 weeks after the last treatment.

Researchers will compare placebo vs. experimental groups to see if psilocybin will increase SVD, and if increases in SVD are associated with cognitive improvements.

DETAILED DESCRIPTION:
The proposed study will investigate the effects of on synaptic vesicular density (SVD) levels as measured by the positron emission tomography (PET) radiotracer, 18F-SynVesT-1, and cognition (i.e., global cognition, executive function, and memory domains) in amnestic Mild Cognitive Impairment (aMCI) and healthy participants. Participants will be randomized to receive either two 25mg doses of psilocybin separated by one week, or two placebo doses separated by one week. Brain scans, clinical, and cognitive assessments will be conducted one week before, and one week, four weeks, and 12 weeks post dosing.

ELIGIBILITY:
Inclusion Criteria

The aMCI participant must meet all of the inclusion criteria to be eligible for this clinical trial:

1. Male or female participants of any race or ethnicity
2. Inpatients or outpatients 60 to 75 years of age (on day of randomization)
3. Diagnosis of MCI based on DSM 5 diagnostic criteria of Minor Neurocognitive Disorder
4. Categorization of episodic memory impairment based on scores ≥ 1.0 SD lower on any of the following measures in comparison to normative data i. Logical Memory Test, ii. California Verbal Learning Test, iii. Brief Visual Memory Test
5. Non-smoker/Non-nicotine user
6. Montreal Cognitive Assessment (MoCA) score = < 26 and MMSE score > = 24
7. Capable of consenting to participate in the research study
8. On a stable dose of medication for at least 2 months [see section 5.6], and unlikely to undergo changes in dose during the study
9. Availability of a study partner who has regular contact with the participant
10. Ability to read and communicate in English (with corrected vision and hearing, if needed)

The Healthy Control participant must meet all of the inclusion criteria to be eligible for this clinical trial:

1. Male or female participants of any race or ethnicity
2. 60 to 75 years of age (on day of randomization)
3. Does not meet SCID-5 criteria for Mild Neurocognitive Disorder, Alzheimer's disease, or other major neurocognitive disorder
4. Non-smoker/Non-nicotine user
5. Capable of consenting to participate in the research study
6. On a stable dose of medication for at least 2 months [see section 5.6], and unlikely to undergo changes in dose during the study
7. Availability of a study partner who has regular contact with the participant
8. Ability to read and communicate in English (with corrected vision and hearing, if needed)

Exclusion Criteria

An individual who meets any of the following criteria will be excluded from participation in this clinical trial:

1. Unwilling or incapable to consent to the study
2. Unstable medical or any concomitant major medical or neurological illness, including presence of a relative or absolute contraindication to psilocybin, i.e. a drug allergy, recent stroke history, uncontrolled hypertension, low or labile blood pressure, recent myocardial infarction, cardiac arrhythmic, severe coronary artery disease, or moderate to severe renal or hepatic impairment.
3. History of head trauma resulting in loss of consciousness > 30 minutes that required medical attention.
4. DSM-5 diagnosis, with active symptoms in the last three months, of major depression; lifetime diagnosis of bipolar disorder; intellectual disability; Alzheimer's Disease; or a psychotic disorder
5. DSM-5 substance dependence (except caffeine) within 12 months of entering the study
6. Anticonvulsant, antidepressant, antipsychotic, mood stabilizer, opioid, or benzodiazepine use
7. Use of serotonergic psychedelic drugs within the past 10 years
8. Positive urine drug screen at the screening visit
9. Having taken a cognitive enhancer (acetylcholinesterase inhibitor or memantine) within the past 6 weeks
10. Acute suicidal or homicidal ideation
11. Receiving treatment with medications such as levetiracetam that blocks SV2a binding, and/or inability to discontinue the following medications before study drug dosing: inhibitors of uridine 5'-diphospho-glucuronosyltransferase (UGT)1A9 and (UGT)1A10, and ALDH inhibitors and alcohol dehydrogenase (ADH) inhibitors.
12. Exceeding allowed annual radiation exposure levels (20 mSv), as outlined by our PET Centre guidelines
13. Having completed multiple PET scans in the past, such that participation in this study would cause participant to exceed lifetime limit (8 PET scans)
14. Metal implants or pacemaker precluding an MRI scan or other contraindications to MRI (e.g., claustrophobia)
15. Female with childbearing potential*, pregnancy (as confirmed by a negative pregnancy test) or breastfeeding
16. Active gender affirming hormonal treatment
17. Any first-degree relative with a diagnosis of schizophrenia-spectrum disorder; psychotic disorder (unless substance-induced or due to a medical condition); or bipolar I or II disorder as determined by the family medical history form and discussions with the participant.
18. Allergies to hydroxypropyl methylcellulose *A woman/female or person who is not of childbearing potential is considered to be postmenopausal after at least 12 months without menstruation. Postmenopausal is defined as 12 consecutive months with no menses without an alternative medical cause. Females/people of childbearing potential are those who have experienced menarche and do not meet the criteria for women not of childbearing potential.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Synaptic Vesicular Density | 3 years
  Synaptic vesicular density will be assessed with PET imaging by measuring the volume of distribution (i.e., defined as the ratio of the radioligand concentration in tissue target region (CT, kBq·cm-3) to that in plasma (CP, kBq·mL-1) at equilibrium) of the [18F]SynVesT-1 radioligand in the cortical and subcortical gray matter regions in the whole brain and more specifically, the hippocampus and dorsolateral prefrontal cortex.

SECONDARY OUTCOMES:
Global Cognition | 3 years
  The results of the neuropsychological battery will be combined to a global cognition composite score as a Z-score, the change of which will be a secondary outcome measure. Z-scores will be comprised of the Mini-Mental State Examination, Montreal Cognitive Assessment, Boston Naming Test, Category Fluency Test, Letter Fluency Test, Trail Making Test Parts A and B, Wisconsin Card Sorting Test, Stroop Neuropsychological Test, Executive Interview, Block Design Test, Clock Drawing Test, Grooved Pegboard, Digit Symbol Test, Logical Memory Test, California Verbal Learning Test, and Modified Rey-Osterrieth Complex Figure, and will be calculated based on the performance of the equated comparison group. Each domain will contribute equally to the global cognition composite score.
Memory | 3 years
  A memory composite Z-score will be generated using the performance on the following individual tests: Logical Memory Test, California Verbal Learning Test, and Modified Rey-Osterrieth Complex Figure. Z-scores will be calculated based on the performance of the equated comparison group, and each domain will contribute equally to the global cognition composite score.
Executive Function | 3 years
  An executive function composite Z-score will be generated using the performance on the following individual tests: Trail Making Test Part B, Wisconsin Card Sorting Test, Stroop Neuropsychological Screening, and the Executive Interview. Z-scores will be calculated based on the performance of the equated comparison group, and each domain will contribute equally to the global cognition composite score.

OTHER OUTCOMES:
Exploratory Cognitive Outcomes | 3 years
  If individual cognitive test scores are significantly different between groups, the mean difference of the individual test scores (i.e., Mini-Mental State Examination, Montreal Cognitive Assessment, Boston Naming Test, Category Fluency Test, Letter Fluency Test, Trail Making Test Parts A and B, Wisconsin Card Sorting Test, Stroop Neuropsychological Test, Executive Interview, Block Design Test, Clock Drawing Test, Grooved Pegboard, Digit Symbol Test, Logical Memory Test, California Verbal Learning Test, and Modified Rey-Osterrieth Complex Figure) will be analyzed separately as exploratory outcomes.
Exploratory Primary and Secondary Outcomes | 3 years
  Primary and secondary outcomes will be compared between aMCI and healthy control groups.
  The means of the primary outcome (i.e., volume of distribution) and secondary outcomes (i.e., cognitive composite Z-scores: global cognition, memory, and executive function) will be compared between aMCI and healthy control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Gerretsen, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Centre for Addiction and Mental Health (CAMH) is the leading mental health and addictions research facility in Canada, and one of the largest in the world. — https://www.camh.ca/en/science-and-research